CLINICAL TRIAL: NCT02637648
Title: Safety and Efficacy of Sodium Oxybate in the Prophylaxis of Headache and Sleep Disturbances in Patients With Chronic and Episodic Cluster Headache
Brief Title: Sodium Oxybate in Patients With Episodic and Chronic Cluster Headache
Acronym: SOinCH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ramin Khatami (Other)
Responsible Party: Sponsor-Investigator, Ramin Khatami, Associative professor, Klinik Barmelweid
Organization: Klinik Barmelweid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BWSO0812
Record Dates: First submitted 2015-12-09; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium oxbate (Experimental): oral administration of sodium oxybate, 6-18ml per night, starting with 6ml in two nightly dosages of 1.5g each, increased by steps of 1.5g every second or third night until treatment response
  Interventions: Drug: Sodium Oxybate
- Placebo (Placebo Comparator): oral administration of placebo, 6-18ml per night, starting with 6ml in two nightly dosages
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Oxybate — parallel Group administration
  Other Names: Xyrem
  Arms: Sodium oxbate
Drug: Placebo — parallel Group administration
  Other Names: not speficied
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effects of sodium oxybate on headache response (frequency), sleep quality and quality of life in the prophylactic treatment of patients with chronic and episodic cluster headache. Oral sodium oxybate, 3-9g per night, starting with 3g in two nightly dosages of 1.5g and increased by steps of 1.5g every second or third night until treatment Response will be evaluated in an interventional, placebo-controlled, double-blind, randomised, parallel group, multicentre study. Primary outcome is reduction of nocturnal pain frequency Secondary outcomes are improvement of sleep quality at a subjective level as assessed by diary and standardized scales (PSQI, FOSQ), duration of pain free episodes, general clinical outcome (global evaluation), clinical global impression (CGI-S, CGI-I, CGI-E), quality of life (SF 36) and daytime sleepiness (Epworth Sleepiness Score).

DETAILED DESCRIPTION:
Multicenter study to test the safety and efficacy of sodium oxybate in the prophylaxis of headache and sleep disturbances in patients with chronic and episodic cluster headache using a placebo-controlled, double blind, randomized study, parallel group design. Patients with predominant nocturnal attacks and poor sleep quality will be evaluated; At least 1 attack every other day and at least 8 attacks cumulatively by the time prior to randomization are required. Sodium oxybate will be orally administered, 3-9g per night, starting with 3g in two nightly dosages of 1.5g (the first at bedtime and the second 4 hours later). Dosage will be gradually increased by steps of 1.5g every second night until treatment response during a titration period of 14 days. Effects od sodium oxybate will be monitored via pain and sleep diaries during a 14 days stable treatment phase by reviewing sleep/pain diaries and Quality of life assessement. Primary outcomes are frequency of nocturnal pain attacks; Main secondary outcomes are frequency, intensity and duration of daytime pain attacks, improvement of sleep quality, quality of life, duration and rates of pain free episodes, decrease in escape medication for acute headache attacks (use of triptans). Safety parameters are ECG, laboratory, depressions scales, vital signs, respiratory polygraphy. Intent-to treat analysis, multivariate analysis of variance (MANOVA) with depending variable (reduction of pain frequency and pain intensity of nocturnal attacks) and the co-variates (age, sex , chronic vs. episodic CH).

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of cluster headache according to the criteria of International Headache Classification (ICHD-II, 2005) of the International Headache Society (IHS).
2. Diagnosis of cluster headache has been made at least 6 weeks after start of screening
3. Patients will have nocturnal pain attacks
4. Duration since onset of current cluster episode at least 1 week
5. Patients will have at least 1 attack per 48 hours and at least 4 attacks cumulatively by the time of visit 2 (prior to randomization)
6. Disturbed sleep quality
7. Patients have expressed a willingness to participate in and complete the study, and signed and dated informed consent prior to beginning protocol required procedures.
8. Women must be surgically sterile or 2 years postmenopausal. Females of child-bearing potential must use a medically accepted effective method of birth control. Patients should agree to continue this method for the duration of the study and for one month after the discontinuation of SO treatment. Women should be negative to serum pregnancy test performed at the screening visit. Females should not be breastfeeding patient.
9. In the opinion of the investigator, the patient must have adequate support to comply with the entire study requirements as described in the protocol (e.g., transportation to and from trial site, self rating scales and diaries completion, drug compliance, scheduled visits, tests).
10. If indicated by investigator, patient must be willing to not operate a car or heavy machinery for 6 hours after the last intake of the investigational drug during the duration of the trial or as long as the investigator deems clinically indicated. In addition, the patient should be willing to abstain during the study any alcohol consumption or behaviours which could interact with the investigational drug.

Exclusion Criteria:

1. The use of sodium oxybate or any previous investigational drugs within 30-day period prior to initial screening visit (V1) for this trial.
2. Change of prophylactic treatment 2 weeks prior of baseline visit 1
3. Have sleep apnea syndrome, defined as an Apnea index > 10 per hour or an Apnea-hypopnea Index (AHI) > 15/h or an oxygen desaturation index (ODI) > 15/h
4. Are taking hypnotics, tranquilizers, antihistamines (except for medication as defined in section 9.4.1. "authorized medication"), benzodiazepines at the start of the baseline period.
5. Patients with psychiatric and neurological disorders, such as moderate or severe psychosis or dementia, bipolar illness, severe anxiety, clinical depression (BDI ≥ 16 with suicidal risk: item G BDI >0).
6. Patients who are experiencing any major illness, including unstable cardiovascular, endocrine, neoplastic, gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurological, pulmonary, and/or renal disease which would place the patient at risk during the trial or compromise the objectives outlined in the protocol.
7. Patients who are unable or unwilling to temporarily discontinue any unauthorized drugs or substances, in particular refrain from alcohol (see section non-authorized treatments).
8. Current or recent (within one year) history of a substance abuse or dependence disorder including alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).
9. Patients taking anticonvulsants are not eligible to participate even if they are willing to washout anticonvulsants for the trial.
10. Patients having other problems that, in the investigators opinion, would preclude the patient's participation and completion of this trial or compromise reliable representation of subjective symptoms.
11. Patients having a history of seizure disorder
12. Patients having a severe renal impairment (e.g. serum creatine greater than 2.0 mg/dl), or a with severe hepatic impairment (abnormal liver function tests SGOT [AST] or SGPT [ALT] more than twice of the upper limit of normal) or elevated serum bilirubin (more than 1.5 times the upper limit of normal) or receiving anti-vitamin K substances.
13. Any significant serious abnormality of the cardiovascular system e.g. recent myocardial infarction, angina, hypertension or dysrhythmias (within the prior 6 months), greater than a first degree AV block.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
nocturnal pain frequency as assessed by patients reports | 4 weeks
  Reduction of nocturnal pain frequency as documented in patients diary,

SECONDARY OUTCOMES:
Improvement of sleep quality | 4 weeks
  Change assessed by PSQI (Pittsburgh Sleep Quality Inventory)
pain free time as assessed by diary | 4 weeks
  number and duration of pain free time periods compared to baseline
Clinical Global Impression | 4 weeks
  Change assessed by CGI-E scale
Quality of life | through study completion
  Assessed by SF 36
Daytime Sleepiness | 4 weeks
  Improvement as assessed by Epworth Sleepiness Score
Escape medication | 4 weeks
  Decrease in escape medication for acute headache attacks (use of triptans)
Depression | 4 weeks
  Change in Beck's depression inventory (BDI-II)
Functional outcome of sleep quality | 4 weeks
  Changes as assessed by questionaire of Functional Outcomes of Sleep Questionaire (FOSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Khatami, MD, Principal Investigator — Clinic Barmelweid AG

REFERENCES:
- [Background] Khatami R, Tartarotti S, Siccoli MM, Bassetti CL, Sandor PS. Long-term efficacy of sodium oxybate in 4 patients with chronic cluster headache. Neurology. 2011 Jul 5;77(1):67-70. doi: 10.1212/WNL.0b013e31822313c6. Epub 2011 May 25. PMID 21613599